CLINICAL TRIAL: NCT00588029
Title: Collection of Tissue, Blood, and Cells to Be Used For Studying the Causes, Prevention, Diagnosis, and Treatment of Breast Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Memorial University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 99-030
Record Dates: First submitted 2007-12-24; First posted 2008-01-08 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Family members
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Cerebro-Spinal Fluid and Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: breast cancer patients
- 2: control subjects without breast cancer

SUMMARY:
The purpose of this study is to collect a blood sample from patients with breast disease (cases) and from individuals without breast cancer (controls)that may be used for research purposes. These blood samples will be used by researchers at Memorial Sloan-Kettering Cancer Center who study the causes of breast cancer, as well as more effective ways to prevent, diagnose, and treat breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* For acquisition of existing breast cancer tissue specimens from the MSKCC Tissue Procurement Service, the only criteria are a pathologically-confirmed diagnosis of invasive breast cancer and the availability of corresponding nonmalignant tissue from each case.
* For the prospective acquisition of blood or saliva from control subjects without breast cancer, eligibility criteria include:
* Any patient with a previous diagnosis of invasive breast cancer who undergoes a palliative procedure related to the presence of a pleural effusion is eligible for the pleural fluid collection aspect of this protocol.
* Any female patient, or any female over the age of 18 accompanying a patient under the care of a physician in the Department of Urology, Department of Surgery, or Department of Medicine.
* Subjects will have no history of preinvasive (carcinoma in situ) or invasive breast cancer.
* Subjects will be eligible without regard to racial, or ethnic status. Attending physicians authorized to obtain informed consent may exercise discretion in excluding individuals for appropriate medical or other (e.g., mentally impaired) reasons.
* For the prospective acquisition of blood, saliva, pleural fluid or cerebrospinal fluid from patients who have or are suspected of having breast cancer or carcinoma in-situ, eligibility criteria include:
* Any patient at MSKCC with a previously confirmed or suspected diagnosis of malignant or premalignant (e.g., carcinoma in situ) breast disease is eligible for inclusion in the blood acquisition aspect of this protocol.
* Any patient with a previous diagnosis of invasive breast cancer who undergoes a palliative procedure related to the presence of a pleural effusion is eligible for the pleural fluid collection aspect of this protocol.
* Any patient with a previous diagnosis of invasive breast cancer with leptomeningeal metastasis who undergoes a routine procedure associated with the collection of cerebrospinal fluid is eligible for the cerebrospinal fluid collection aspect of this protocol.
* All subjects must be under the care of one or more members of the MSKCC Breast Disease Management Team at the time of enrollment.
* Subjects may have received prior hormonal therapy, cytotoxic chemotherapy, radiation therapy, or surgical therapy at MSKCC or another institution.
* All subjects must be 18 years or older
* Subjects will be eligible without regard to sex, racial, or ethnic status. It is anticipated that approximately 99% of the patients will be female. Attending physicians authorized to obtain informed consent may exercise discretion in excluding individuals for appropriate medical or other (e.g., mentally impaired) reasons.
* If, after pathologic diagnosis, preinvasive or invasive breast disease is not found, patients previously consented for the blood collection aspect of this protocol will not be included.

Exclusion Criteria:

* For the prospective acquisition of blood or saliva from control subjects without breast cancer, ineligibility criteria include:

  * A first degree relative (mother, daughter, sister, father, brother or son) who has been diagnosed with breast cancer.
  * A personal history of breast cancer, lobular carcinoma in situ or atypia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients seen at Memorial Sloan-Kettering Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 1999-07; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
None. This is a tissue banking study. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mark Robson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan-Kettering Cancer, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm